CLINICAL TRIAL: NCT00004795
Title: Phase II/III Randomized, Double-Blind, Placebo-Controlled Study of Dehydroepiandrosterone in Women With Mild to Moderate Systemic Lupus Erythematosus
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Northwestern University (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: 199/11930; NU-517
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-12

CONDITIONS: Systemic Lupus Erythematosus
Keywords: arthritis & connective tissue diseases; immunologic disorders and infectious disorders; rare disease; systemic lupus erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Arthritis; Connective Tissue Diseases; Immune System Diseases; Communicable Diseases; Rare Diseases | interventions — Dehydroepiandrosterone

INTERVENTIONS:
Drug: dehydroepiandrosterone

SUMMARY:
OBJECTIVES: I. Evaluate the safety and efficacy of synthetic dehydroepiandrosterone (GL701) in women with prednisone-dependent systemic lupus erythematosus.

II. Describe the pharmacokinetics of GL701.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, double-blind study. Patients are stratified by participating institution.

Patients are randomly assigned to 1 of 2 doses of oral dehydroepiandrosterone or placebo, administered daily for a minimum of 7 months. A prednisone taper is attempted each month in patients with stable or improving disease. Therapy continues until a successful prednisone taper is achieved and sustained for at least 2 months, or until a maximum of 9 months.

Patients are followed for 1 year after entry.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Systemic lupus erythematosus by American College of Rheumatology criteria Mild to moderate disease characterized as follows: Prednisone dose (or equivalent) 10 to 30 mg/day No daily dose 1 mg/kg or greater No alternate-day regimen Failed prednisone taper in last 12 months and dose stable for at least 6 weeks prior to entry OR No attempt to taper in last 12 months and dose stable for at least 3 months prior to entry No prior participation in double-blind dehydroepiandrosterone (DHEA) study at Stanford University --Prior/Concurrent Therapy-- No concurrent immunosuppressants No concurrent participation in other clinical studies No investigational agents within the longer of 30 days or 10 half lives of the agent At least 3 months since the following: Adrenocorticotropin hormone Androgens Cyclophosphamide Azathioprine Intravenous immune globulin Other immunosuppressants At least 1 month since any change in dose of concurrent nonsteroidal anti- inflammatory drugs or hydroxychloroquine --Patient Characteristics-- No hypersensitivity to DHEA or inactive ingredient in DHEA, i.e.: Cornstarch Lactose Magnesium stearate No condition that would prevent adequate compliance with study No history of breast cancer or reproductive tract malignancy Negative pregnancy test required within 2 weeks prior to entry Reliable contraception required of fertile women No estrogen-containing oral contraceptive

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190
Dates: Start 1994-08

CONTACTS AND LOCATIONS:
Overall Officials: Rosalind Ramsey-Goldman, Study Chair — Northwestern University